CLINICAL TRIAL: NCT01144091
Title: Renal Effect of Pentoxyphylline in High Risk Patients Undergoing Angiography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMC10059-2010
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2012-09

CONDITIONS: Contrast Induced Nephropathy; Diabetes Mellitus
Keywords: diabetes mellitus; creatinin level; contrast induced nephropathy; prevention contrast induced nephropathy in high risk patients
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- pentoxyphylline cardio (Experimental): Patients with chronic renal failure (CRF) and/or diabetes mellitus (DM) who are about to go to undergo coronary angiography
  Interventions: Drug: pentoxyphylline
- placebo cardio (Placebo Comparator): Patients with chronic renal failure (CRF) and/or diabetes mellitus (DM) who are about to go to undergo coronary angiography
  Interventions: Drug: placebo
- radiology pentoxyphylline (Experimental): Patients with chronic renal failure (CRF) and/or diabetes mellitus (DM) who are about to go to undergo computed tomography with contrast
  Interventions: Drug: pentoxiphylline
- radiology placebo (Placebo Comparator): Patients with chronic renal failure (CRF) and/or diabetes mellitus (DM) who are about to go to undergo computed tomography with contrast
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pentoxyphylline — pentoxyphylline tablets, 400 mg per tablet, 3 times a day one day before, on the day of the procedure and for another 48 hours.
  Other Names: Oxopurin; Trental; Pentoxifylline-Teva
  Arms: pentoxyphylline cardio
Drug: placebo — placebo tablets 3 times a day one day before, on the day of the procedure and for another 48 hours.
  Arms: placebo cardio
Drug: pentoxiphylline — pentoxyphylline tablets, 400 mg per tablet, 3 times a day one day before, on the day of the procedure and for another 48 hours.
  Other Names: terental; oxopurin; Pentoxifylline-Teva
  Arms: radiology pentoxyphylline
Drug: placebo — placebo tablets 3 times a day one day before, on the day of the procedure and for another 48 hours.
  Arms: radiology placebo

SUMMARY:
The investigators will study 2 separate groups:

* Cardiology patients undergoing invasive coronary angiography +/- PCI (Percutaneous coronary intervention).
* Patients undergoing CT examination with contrast medium. All patients will receive intravenous (I.V) hydration for 8-12h before and 36 to 48 h after angiography with 0.45% saline 100ml/h.

All patients will receive oral N-acetyl cysteine 1200 mg twice daily, a day before, on the day of the angiography and for another 48 hours.

In addition, patients will be assigned to receive oral pentoxyphylline (P group) or placebo (C - control group) tablets 3 times a day one day before, on the day of the procedure and for another 48 hours.

Baseline Serum Creatinine (S.Cr) levels in will be taken before angiography and two days after angiography. Radio-contrast nephropathy is defined, in this study, as increase in serum ≥ 25 % of baseline after injection of the radio-contrast agent. Pentoxyfylline is an orally active haemorheological agent for the treatment of peripheral vascular disease, cerebrovascular disease and a number of other conditions involving a defective regional microcirculation. Pentoxyfylline acts primarily by increasing red blood cell deformability, by reducing blood viscosity and by decreasing the potential for platelet aggregation and thrombus formation (mechanism unclear). Pentoxyfylline has also proven to have a significant anti inflammatory effect as well as anti oxidant effect, mechanisms considered to be important patho-physiological causes of contrast induced nephropathy.

DETAILED DESCRIPTION:
Impairment of renal function following exposure to intravenous radio-graphic contrast materials is the third major cause of renal hospital acquired renal dysfunction. Renal dysfunction occurs most often in patients with chronic renal failure and or patients with diabetes mellitus and contributes to the morbidity and mortality. Previous research work proved that the use volume expansion with N-acetyl cysteine (NAC) is superior to volume expiation alone to prevent renal impairment due to radio-contrast5. NAC a potent anti oxidant may prevent CIN by stopping direct oxidative tissue damage and by improving renal hemodynamics.Pentoxyfylline has also proven to have a significant anti inflammatory effect as well as anti oxidant effect.Preangiographic and the highest post-angiographic values of Creatinine and eGFR (estimated glomerular filtration rate) will be recorded. Levels of the biomarker Neutrophil - gelatinase - associated lipocalin (NGAL) will be tested randomly in 49 patients p as a biomarker for contrast induced nephropathy. Blood serology for NGAL will be drown from patients before the procedure and 2 hours after angiography.

ELIGIBILITY:
Inclusion Criteria:

Cardiology patients:

1. Hospitalization for ACS (acute coronary syndrome) with NSTEMI or Unstable Angina
2. Diabetic patients (treated with insulin or oral hypoglycemic drugs) or patients with basal serum creatinine greater than 1.3mg/dl in females and 1.5 mg/dl in male patients.
3. Informed consent
4. Age between 18-75

Radiology patients:

1. Radiology patients should be diabetic patients (treated with insulin or oral hypoglycemic drugs) or patients with basal serum creatinine of 1.3mg/dl in females and 1.5 mg/dl in male patients.
2. Informed consent
3. Age between 18-75

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-04 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The purpose of the study is to examine the potential renal protective effect of pentoxyphylline in high-risk patients undergoing angiography | one year
  The difference between preangiographic and postangiographic values (∆) for S.Cr and eGFR will be calculated and compared between groups. Baseline Serum Creatinine (S.Cr) levels in will be taken before angiography and levels of the biomarker Neutrophil - gelatinase - associated lipocalin (NGAL) will be tested randomly in 49 patients.contrast induced nephropathy.
  Comparison of the ∆ between the preangiographic and postangiographic values for S.Cr and eGFR will be performed between the groups.

SECONDARY OUTCOMES:
The purpose of the study is to examine the potential renal protective effect of pentoxyphylline in diabetic patients undergoing angiography | one year
  Subgroup analysis will be performed for subgroups of patients with diabetes mellitus (DM)
The purpose of the study is to examine the potential renal protective effect of pentoxyphylline in patients with elevated base line creatinin level > 2 undergoing angiography | one year
  Subgroup analysis will be performed for subgroups of patients high S.Cr levels before the procedure